CLINICAL TRIAL: NCT01916954
Title: Comparison of Two Regimens of Artemether-lumefantrine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Pregnant Women in the Democratic Republic of Congo
Brief Title: Comparison of Two Regimens of Artemether-lumefantrine for the Treatment of Malaria in Pregnancy
Acronym: ALN5P
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Kinshasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALN5P
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Malaria
Keywords: Malaria; Pregnancy; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-day artemether-lumefantrine (Active Comparator): Standard artemether-lumefantrine regimen (3-day treatment)
  Interventions: Drug: 3-day artemether-lumefantrine
- 5-day artemether-lumefantrine (Experimental): Artemether-lumefantrine extended regimen (5-day treatment)
  Interventions: Drug: 5-day artemether-lumefantrine

INTERVENTIONS:
Drug: 3-day artemether-lumefantrine
  Arms: 3-day artemether-lumefantrine
Drug: 5-day artemether-lumefantrine
  Arms: 5-day artemether-lumefantrine

SUMMARY:
Malaria in pregnancy is a major cause of maternal and newborn morbidity and mortality in sub-Saharan Africa]. Effective antimalarial preventive and treatment regimens can significantly reduce malaria-related morbidity and mortality in the mother and baby. However, therapeutic choices are limited by concerns about possible toxicity to the fetus and because of these concerns pregnant women are normally excluded from clinical trials. This, combined with the lack of adverse events reporting system, results in a scarcity of data on drug safety and efficacy in pregnancy. Moreover, changes in the maternal physiology in pregnancy often alter the pharmacokinetic of drugs. Artemether-lumefantrine (ALN) is a highly efficacious artemisinin-based combination therapy approved by the World Health Organisation for use in the 2nd and 3rd trimesters, although it is still infrequently used in pregnancy and there is uncertainty as to the optimum dose. The pharmacokinetics of ALN are altered in pregnancy, resulting in reduced plasma concentrations and while the standard adult dose is still effective in high transmission settings, where pregnant women have higher levels of immunity, efficacy is reduced significantly in low transmission settings where women have lower levels of immunity. Inadequate antimalarial treatment dosing in pregnancy risks treatment failure or breakthrough infection and exposure of malaria parasites to sub-therapeutic drug concentrations thus selecting for drug resistance.

DETAILED DESCRIPTION:
The aim of the current trial is to compare the standard 3-day regimen of artemether-lumefantrine to a 5-day regimen of artemether-lumefantrine in a group of pregnant women and a control of non-pregnant women with uncomplicated P. falciparum malaria. The pharmacokinetics of lumefantrine is modified in pregnancy and the standard regimen used for treatment of adults might not be sufficient to cure malaria, therefore exposing pregnant women to sub-therapeutic drug levels and increased risk of clinical failure. Previous pharmacokinetic studies have shown that the standard 3-day treatment during pregnancy results in reduced plasma concentrations of artemether, dihydroartemisinin and lumefantrine and a faster elimination of lumefantrine. Low lumefantrine plasma concentrations at day 7 are associated with therapeutic failure. Population-based simulations suggest that increased dose and treatment duration are needed for adequate drug exposure in these patients. We propose to assess the pharmacokinetics of a longer regimen of artemether-lumefantrine, (10 doses of artemether-lumefantrine over five days) compared to the standard regimen, (6 doses of artemether-lumefantrine over three days) in a small group of pregnant African women with uncomplicated P. falciparum malaria. The longer regimen should ensure that curative plasma concentration of lumefantrine is reached, and is unlikely to result in any increased frequency of adverse events.

ELIGIBILITY:
Inclusion criteria for non pregnant women:

* Age ≥18 and ≤ 45 years
* P. falciparum parasitemia ≥ 100 parasites/μL and less than 200.000 parasites/μL
* Hematocrit ≥21%
* Negative HIV test
* Negative pregnancy test*
* Written informed consent provided
* Willing to stay for 3 or 5 days at the hospital and to comply with the follow-up schedule

Inclusion criteria for pregnant women (in addition to the above criteria except*):

* Gestational Age ≥ 14 weeks confirmed by ultrasound
* Singleton viable fetus

Exclusion criteria for non-pregnant women:

* Severe malaria or signs of severe malaria
* Medical conditions requiring concomitant drug treatment or transfer to a different hospital
* Intake of artemether-lumefantrine within the two previous 2 weeks
* Known allergy to the study drugs
* Previous participation in this study or current participation in other studies

Exclusion criteria for pregnant women (in addition to the above criteria):

* Signs of labour
* Fetal abnormalities identified by ultrasound

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics measures | 1 year
  Drug plasma concentration profiles for lumefantrine, artemether and dihydroartemisinin will be characterized for each patient. Ten samples per patient will be taken at fixed and random times.

SECONDARY OUTCOMES:
Tolerability and safety measures | 2 years
  Detection and assessment of adverse events during the therapy and in the follow-up period.

OTHER OUTCOMES:
Efficacy measures | 1 year
  Therapeutic efficacy of the treatment will be assessed in the follow-up period according to WHO protocol for the evaluation of antimalarial efficacy. Therapeutic responses will be correlated with drug concentration profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas P Day, MD PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Kinshasa, Democratic Republic of Congo, Kinshasa, Republic of the Congo

REFERENCES:
- [Derived] Onyamboko MA, Hoglund RM, Lee SJ, Kabedi C, Kayembe D, Badjanga BB, Turner GDH, Jackson NV, Tarning J, McGready R, Nosten F, White NJ, Day NPJ, Fanello C. A Randomized Controlled Trial of Three- versus Five-Day Artemether-Lumefantrine Regimens for Treatment of Uncomplicated Plasmodium falciparum Malaria in Pregnancy in Africa. Antimicrob Agents Chemother. 2020 Feb 21;64(3):e01140-19. doi: 10.1128/AAC.01140-19. Print 2020 Feb 21. PMID 31818818